CLINICAL TRIAL: NCT04684147
Title: Phase Ⅱ Clinical Trial of CNCT19 Cell Injection in the Treatment of CD19 Positive Relapsed or Refractory Acute Lymphoblastic Leukemia
Brief Title: Clinical Trial of CNCT19 Cell Injection in the Treatment of Relapsed or Refractory Acute Lymphoblastic Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Juventas Cell Therapy Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HY001201
Record Dates: First submitted 2020-12-09; First posted 2020-12-24 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Relapsed or Refractory Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Recurrence; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single dose of CNCT19 (Experimental): A conditioning chemotherapy regimen of fludarabine and cyclophosphamide will be administered followed by investigational treatment, CNCT19.
  Interventions: Biological: single dose of CNCT19

INTERVENTIONS:
Biological: single dose of CNCT19 — Dose: 0.5 x 10^8 CNCT19 Cell Injection via intravenous infusion. Drug: Fludarabine Drug: Cyclophosphamide

SUMMARY:
The study is a Phase II, single-arm, open-label, single-dose clinical trial, and its primary objective is to evaluate the efficacy and safety of CNCT19 Cell Injection in the treatment of CD19 positive Relapsed or Refractory acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
The study is a Phase II, single-arm, open-label, single-dose clinical trial, and its primary objective is to evaluate the efficacy and safety of CNCT19 Cell Injection in the treatment of CD19 positive Relapsed or Refractory acute lymphoblastic leukemia. The study consists of screening period (8 weeks), treatment period (4 weeks), and follow-up period (2 years at most).

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent is signed by the subject.
2. Age 18 to 65.
3. Relapsed or refractory acute lymphoblastic leukemia (ALL). (1) Relapse within 12 months of first remission; (2)a. Without remission after more than 6 weeks of induction chemotherapy or without remission after 2 cycles of induction chemotherapy regimen; c. 2nd or greater Bone Marrow (BM) relapse OR; d. First relapse after chemotherapy, without remission after at least 1 rescue treatment; e. Any BM relapse after autologous or allogeneic stem cell transplantation (SCT).
4. Documentation of CD19 tumor expression demonstrated in bone marrow or peripheral blood within 3 months of study entry.
5. Patients with Philadelphia chromosome positive (Ph+) ALL are eligible if they are intolerant to or have failed 2 generation of tyrosine kinase inhibitor therapy (TKI); no TKI salvage treatments if the patient has a T315I mutation.
6. Bone marrow with ≥ 5% lymphoblasts by morphologic assessment at screening.
7. Eastern cooperative oncology group (ECOG) performance status of 0 to 1.
8. Adequate organ function defined as:

   1. aspartate aminotransferase (AST) ≤ 3 upper limit of normal (ULN);
   2. Serum alanine aminotransferase (ALT) ≤ 3 upper limit of normal (ULN);
   3. Total bilirubin ≤ 2 ULN, except in individuals with Gilbert's syndrome; Note: Patients with Gilbert's syndrome that bilirubin ≤ 3 ULN and direct bilirubin ≤ 1.5 ULN will be eligible;
   4. A serum creatinine≤ 1.5 ULN or Creatine removal rate ≥ 60mL/min (Cockcroft and Gault）;
   5. Must have a minimum level of pulmonary reserve as ≤ Grade 1 dyspnea and oxygen saturation > 91% on room air;
   6. International normalized ratio (INR) ≤ 1.5 ULN and activated partial thromboplastin time (APTT) ≤ 1.5 ULN.
9. Vascular conditions for apheresis.
10. Women of childbearing age have a negative blood / urine pregnancy test within 3 days before apheresis and the CNCT19 infusion. Women of child-bearing potential and all male participants must use highly effective methods of contraception throughout the study and for a period of at least two years after the CNCT19 infusion.

Exclusion Criteria:

1. Active Central Nervous System (CNS) involvement by malignancy.
2. Isolated extra-medullary disease relapse.
3. Patients who received chemotherapy within 2 weeks before CNCT19 infusion. The following situations are excluded:

   1. Lymphodepleting Chemotherapy prescribed by the protocol;
   2. Tyrosine kinase inhibitors (TKI) and hydroxyurea must be stopped > 72 hours prior to CNCT19 infusion;
   3. The following drugs must be stopped > 1 week prior to CNCT19 infusion: 6-mercaptopurine, 6-thioguanine, methotrexate (<25 mg / m2), cytosine arabinoside (<100 mg / m2 / d), vincristine, asparaginase;
   4. CNS prophylaxis treatment must be stopped > 1 week prior to CNCT19 infusion;
   5. Pegylated-asparaginase must be stopped > 4 weeks prior to CNCT19 infusion.
4. Radiotherapy before CNCT19 infusion:

   Non-CNS site of radiation completed < 2 weeks prior to CNCT19 Infusion; CNS directed radiation completed < 8 weeks prior to CNCT19 infusion.
5. Therapeutic systemic doses of steroids were stopped < 72 hours prior to CNCT19 infusion. However, the following physiological replacement doses of steroids are allowed: < 10 mg/day hydrocortisone or equivalent.
6. Has received anthracycline/anthraquinone drug treatment exceeding the maximum cumulative dose recommended by the guidelines, estimated by investigators before screening, as follows:

   * Doxorubicin: 550mg/m2 (radiotherapy or combined medication, <(radiotherapy or combined medication, <350~400 mg/m2);
   * Epirubicin: 900~1000 mg/m2 (Adriamycin used, <800 mg/m2);
   * Pirarubicin: 950 mg/m2;
   * Daunorubicin: 550 mg/m2;
   * Demethoxydaunorubicin: 290 mg/m2;
   * Aclarithromycin: 2000 mg/m2 (Adriamycin used, <800 mg/m2);
   * Mitoxantrone: 160 mg/m2 (using doxorubicin, <120 mg/m2);
7. Has had treatment with any prior CAR-T therapy.
8. Patients with acute graft-versus-host disease (GVHD) or moderate-to-severe chronic GVHD within 4 weeks before screening; Patients who have received systemic drug therapy for GVHD within 4 weeks before CNCT19 infusion.
9. Patients with systemic vasculitis.
10. Patients complying with any of hepatitis B surface antigen (HBsAg) and/or hepatitis B e antigen (HBeAg) positive, hepatitis B e antibody (HBe-Ab) and/or hepatitis B core antibody (HBc-Ab) positive and HBV-DNA copies being more than the lower limit of detection, hepatitis C antibody (HCV-Ab) positive, anti-treponemia pallidum antibody (TP-Ab) positive, EBV-DNA, and CMV-DNA copies being more than the lower limit of detection.
11. Prior malignancy. Patients with Prior malignancy that has been cured for ≥ 5 years or has a low risk of relapse, judged by investigators are excluded.
12. a. Left Ventricular Ejection Fraction (LVEF) ≤45%; b. III/IV congestive heart failure (NYHA); c. Severe arrhythmia, or clinically significant conduction abnormalities that can be seen on ECG, including QTc interval ≥480ms (QTcB=QT/RR1/2); d. Hypertension that has not been controlled after standard treatment (systolic ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg); e. Unstable angina; f. Myocardial infarction or Coronary Artery Bypass Graft Surgery, heart stent surgery < 6 months prior to CNCT19 infusion; f. Clinically significant valvular disease; g. Other heart diseases that have been judged by the investigator to be unsuitable for receiving cell therapy.
13. Clinically significant pleural effusion.
14. Patients with a history of epilepsy, cerebrovascular ischemia / hemorrhage, cerebellar disease or other active central nervous system diseases.
15. History of deep vein thrombosis or pulmonary embolism within 6 months of screening.
16. Known history of hypersensitivity to ingredients used in the drug.
17. Has had treat with live vaccine within 6 weeks prior to screening.
18. Patients with active infections in screening.
19. Life expectancy < 3 months.
20. Patient in other interventional clinical studies, who received live investigational product, including: Unlisted new drugs within 3 months before CNCT19 injection, marketed drug within 5 half-lives before CNCT19 injection, or who intend to participate in another clinical trial or receive anti-tumor therapy outside the protocol during the entire study.
21. Patients with other conditions making the patients unsuitable for receiving cell therapy as judged by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-12-24 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Remission Rate (ORR), which includes Complete Remission (CR) and Complete Remission with Incomplete Blood Count Recovery (CRi) as determined by Independent Review Committee (IRC). | At 3 months after infusion
  The Investigators' evaluation results of ORR will be subjected to sensitivity analysis.

SECONDARY OUTCOMES:
Overall Remission Rate (ORR) with minimal residual disease (MRD) negative bone marrow as determined by IRC and Investigators. | 3 months
  MRD negative status as determined using flow cytometry.
Overall Remission Rate (ORR) as determined by IRC and Investigators. | 28 days
  The proportion of patients who have achieved CR or CRi.
Overall Remission Rate (ORR) with minimal residual disease (MRD) negative bone marrow as determined by IRC and Investigators. | 28 days
  MRD negative status as determined using flow cytometry.
Relapse Free Survival (RFS) as determined by IRC and Investigators. | 2 years
  RFS means the duration from reaching the response CR or CRi to the first defined relapse, or death due to any cause, whichever comes first.
Event free survival (EFS) as determined by IRC and Investigators. | 2 years
  EFS means duration from the CNCT19 Cell Injection infusion to death for any reason after remission, relapse, treatment failure, no response, or termination (because of death, adverse event, lack of efficacy, progression, new anti-tumor treatments.
Duration of remission (DOR) as determined by IRC and Investigators. | 2 years
  DOR means the duration from reaching the response CR or CRi to the first defined relapse, or death due to any cause, whichever comes first.
Best overall response (BOR) as determined by IRC and Investigators. | 2 years
  The proportion of patients who have achieved the best effect (CR or CRi) after the experimental treatment.
Overall survival (OS) as determined by IRC and Investigators. | 2 years
  OS is defined as the time from the CNCT19 Cell Injection infusion to the date of death due to any cause.
In vivo cellular Pharmacokinetic (PK) profile of CNCT19 in units of transgene copy number per genomic DNA (gDNA) amount. | 2 years
  Characterize the pharmacokinetic (PK) profile in blood, bone marrow (if available) and Cerebral Spinal Fluid (CSF) (if available) by qPCR.
In vivo cellular Pharmacokinetic (PK) profile of CNCT19 in units of percent of CAR-positive cells. | 2 years
  Characterize the pharmacokinetic (PK) profile in blood, bone marrow (if available) and Cerebral Spinal Fluid (CSF) (if available) by Flow Cytometry.
Concentration of Cytokines in Serum. | 28 days
  Collected as pharmacodynamic data, including IL-6 at list.
Concentration of ferritin in Serum. | 28 days
  Collected as pharmacodynamic data.
Concentration of C reactive protein in serum. | 28 days
  Collected as pharmacodynamic data.
Prevalence and incidence of humoral immunogenicity (anti-drug antibodies) to CNCT19. | 2 years
  Collected as Immunogenicity data.

CONTACTS AND LOCATIONS:
Overall Officials: Jianxiang Wang, Dr., Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (11):
- China (11):
  - Beijing Boren Hospital, Beijing, Beijing Municipality
  - Xinqiao Hospital of TMMU, Chongqing, Chongqing Municipality
  - Nanfang Hospital, Guangzhou, Guangdong
  - Yanda hospital, Hebei medical university, Sanhe, Hebei
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - The affiliated hospital of Xuzhou medical university, Xuzhou, Jiangsu
  - Tongji Hospital of Tongji University, Shanghai, Shanghai Municipality
  - West China Hospital，Sichuan University, Chengdu, Sichuan
  - Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University school of Medicine, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Wang Y, Lv L, Song Y, Wei X, Zhou H, Liu Q, Xu K, Yan D, Zhang C, Liu S, Jin J, Mei H, Niu T, Liang A, Gu R, Ren J, Feng Y, Jin W, Zhou Y, Deng Y, Wang J. Inaticabtagene autoleucel in adult relapsed or refractory B-cell acute lymphoblastic leukemia. Blood Adv. 2025 Feb 25;9(4):836-843. doi: 10.1182/bloodadvances.2024014182. PMID 39626300
- [Derived] Shi Z, Zhu Y, Zhang J, Chen B. Monoclonal antibodies: new chance in the management of B-cell acute lymphoblastic leukemia. Hematology. 2022 Dec;27(1):642-652. doi: 10.1080/16078454.2022.2074704. PMID 35622074